CLINICAL TRIAL: NCT01275118
Title: Comparative Study of Photopic and Mesopic Distance, Intermediate and Near Visual Acuity, and Spectacle Independence With Bilateral Implantation of the Tecnis Multifocal (TMF) Intraocular Lens or Crystalens AO (CAO) Intraocular Lens
Brief Title: Comparison of Postoperative Visual Acuity and Spectacle Independence Between the Tecnis Multifocal Intraoculer Lens (IOL) and the Crystalens Accommodating IOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mark Packer, MD, FACS (Other)
Collaborators: Abbott Medical Optics (Industry)
Responsible Party: Sponsor-Investigator, Mark Packer, MD, FACS, Sponsor-Investigator, Drs. Fine, Hoffman and Packer, LLC
Organization: Drs. Fine, Hoffman and Packer, LLC (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMF-09-002 Rev.5
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Tecnis Multifocal IOL — Presbyopia correcting IOL
Device: crystalens Accommodating IOL — Presbyopia correcting IOL

SUMMARY:
Comparison of postoperative visual acuity and spectacle independence between the Tecnis Multifocal Intraoculer Lens (IOL) and the crystalens Accommodating IOL

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Status post bilateral cataract or refractive lens surgery (with or without LRI) and implantation of Tecnis™ Multifocal IOL or Crystalens™ AO Accommodating IOL
* Best-corrected ETDRS equivalent visual acuity of 20/30 or better in each eye
* Naturally dilated pupil size (in dim light) > 3.5 mm (with no dilation medications) for both eyes
* Clear intraocular media (no posterior capsular opacification, or status post YAG capsulotomy)
* Availability, willingness, and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

* Ocular disease which could potentially limit uncorrected visual acuity or visual performance.
* Use of systemic or ocular medications that may affect visual outcomes
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus, immunocompromised, etc.)
* Uncontrolled systemic or ocular disease
* History of ocular trauma
* History of ocular surgery other than that required for inclusion in this study
* Amblyopia or strabismus
* Known pathology that may affect visual acuity; particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.)
* Diagnosed degenerative visual disorders (e.g. macular degeneration, or other retinal disorders) that are predicted to cause future acuity losses to a level of worse than 20/30
* Subjects who may be expected to require retinal laser treatment or other surgical intervention
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome)
* Pupil abnormalities (non-reactive, tonic pupils or abnormally shaped pupils)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Visual function | 3 months postoperatively

SECONDARY OUTCOMES:
Use of spectacle correction and vision-related quality of life | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Mark Packer, MD, FACS, CPI, Principal Investigator — Drs. Fine, Hoffman and Packer, LLC
Locations (1):
- Drs. Fine, Hoffman and Packer, LLC, Eugene, Oregon, United States